CLINICAL TRIAL: NCT02973893
Title: A Prospective, Multi-Center, Double-Blind, Randomized, Placebo-Controlled Trial Comparing Two Doses of VF001-DP to Placebo as an Adjunct to Standard Care in Patients With Chronic Venous Leg Ulcers
Brief Title: Study of VF001-DP in Patients With Chronic Venous Leg Ulcers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Factor Therapeutics Ltd. (Industry)
Collaborators: Parexel (Industry); ARANZ Medical (Other); ALMAC Clinical Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VF00102
Record Dates: First submitted 2016-11-07; First posted 2016-11-25 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Ulcer; Leg Ulcer; Varicose Ulcer; Pathologic Processes; Skin Ulcer; Skin Diseases; Vascular Diseases; Cardiovascular Diseases
Keywords: Chronic Venous Leg Ulcer
MeSH Terms: conditions — Ulcer; Leg Ulcer; Varicose Ulcer; Pathologic Processes; Skin Ulcer; Skin Diseases; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo plus Standard Care (Placebo Comparator): Placebo plus Standard Care
  Interventions: Biological: Placebo
- VF001-DP LD plus Standard Care (Experimental): VF001-DP (14 micrograms per treatment) and Standard Care (low dose [LD])
  Interventions: Biological: VF001-DP LD
- VF001-DP HD plus Standard Care (Experimental): VF001-DP (140 micrograms per treatment) and Standard Care (high dose [HD])
  Interventions: Biological: VF001-DP HD

INTERVENTIONS:
Biological: Placebo — Placebo
  Arms: Placebo plus Standard Care
Biological: VF001-DP LD — VF001-DP contains parts of normal vitronectin and Insulin-like growth factor 1 (IGF-I) combined in a single protein.
  Arms: VF001-DP LD plus Standard Care
Biological: VF001-DP HD — VF001-DP contains parts of normal vitronectin and Insulin-like growth factor 1 (IGF-I) combined in a single protein.
  Arms: VF001-DP HD plus Standard Care

SUMMARY:
The purpose of this study is to determine if VF001-DP improves wound healing in chronic venous leg ulcers compared to standard care only.

DETAILED DESCRIPTION:
Objective: The objective of this study is to demonstrate the effectiveness and safety of VF001-DP as an adjunct to standard care (SC) in the treatment of chronic venous leg ulcers (VLUs) compared to Placebo with SC over the course of the 12-week Treatment Phase.

Design: This study is a multi-center, randomized, double-blind, placebo-controlled dose-response study designed to evaluate VF-001-DP as an adjunct to SC, versus Placebo and SC in the treatment of chronic VLUs. The SC therapy for VLUs is a moisture retentive ulcer dressing and multi-layer compression therapy. Mepitel® and Coban2® have been chosen to be used as SC in this trial.

The study will have three (3) phases: Screening (2 weeks), Treatment Phase (12 weeks) and Follow-Up (12 weeks).

Only patients whose study ulcer does not exhibit more than 30% change (increase or decrease) in ulcer size post-debridement between Screening Phase Visit (S1) and Treatment Phase Visit (T1) and who continue to meet eligibility criteria at T1 will be randomized to receive either the Active Treatment group (VF001-DP low or high dose plus SC) or the Control Treatment group (Placebo plus SC) in a ratio of 1:1:1.

Treatment: Eligible patients will be assigned to one of the following treatment groups:

* Placebo and SC
* VF001-DP (14 micrograms per treatment) and SC (low dose [LD])
* VF001-DP (140 micrograms per treatment) and SC (high dose [HD]).

The investigational product (IP), i.e., VF001-DP and placebo, will be supplied in 1 mL syringes each containing 0.5 mL of either VF001-DP or Placebo.

The IP contains parts of normal vitronectin and Insulin-like growth factor 1 (IGF-I) combined in a single protein (vitronectin, amino acids 1-64 of the human sequence and IGF-I amino acids 1-70 of the human sequence), 14 μg or 140 μg protein in 0.5 mL of Phosphate Buffered Saline, pH 7.2. VF001-DP is manufactured utilizing an expression vector system in yeast to Good Manufacturing Practice (GMP) and is not made with and does not include any products of human or animal origin.

Number of Patients: It is planned to recruit 168 patients (56 per treatment group) at 26 centres in USA for this study.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Ankle-Brachial Pressure Index (ABI) ≥0.80. (Calculations will be made using measurements from both posterior tibial and dorsalis pedis arteries as well as both arms).
3. Presence of VLUs extending through the full thickness of the skin but not down to muscle, tendon or bone. In the case of more than one ulcer, the largest ulcer (compliant with study criteria) will be chosen as the study ulcer and treated in the study. Other ulcerations, if present on the same leg must be at least 2 cm apart from the study ulcer.
4. Venous disease confirmed by Doppler ultrasonography to demonstrate reflux of >0.5 seconds in saphenous (great or small), calf perforators or the deep venous system. Patients with prior venous surgery (i.e., varicose vein stripping, endovenous ablation) may be included if they still demonstrate significant reflux in a remaining venous segment and the ulcer continues to suffer poor healing because of venous hypertension.
5. Ulcer which has been present and treated with standard care (moisture retentive ulcer dressings and compression bandaging not limited to Mepitel® and Coban2®) for at least one month prior to the initial Screening Visit.
6. Moderate severity ulcer at the T1 visit (post-debridement) complying with the following requirements of the Margolis Predictive Score Baseline Wound Area and Wound Duration:

   1. 1(a) 2.5 cm2 to not-more-than 5 cm2 and not-less-than 6 months or;
   2. 1(b) Not-less-than 5 cm2 to not-more-than 15 cm2 and not-more-than 6 months
7. Ulcer with a clean, granulating base free of adherent slough at the T1 visit (post-debridement).
8. Female patients of childbearing potential, willing to use acceptable methods of contraception (birth control pills, barriers, or sexual abstinence). A urine pregnancy test must be performed, and negative at the T1 visit.
9. Patient able to understand the study procedures and willing to participate in the clinical study and able to comply with study visit schedule.
10. Provide signed informed consent.

Exclusion Criteria

1. Ulcer(s) deemed by the Investigator to be caused by a medical condition other than venous insufficiency. These may include, but are not limited to: fungal ulcerations, malignant ulcerations, diabetic (neuropathic) ulcerations, and ulcerations due to arterial insufficiency.
2. Increase or decrease by >30% in the study ulcer surface area at the T1 visit post-debridement as compared to the S1 visit study ulcer surface area post-debridement.
3. Ulcer exhibits clinical signs and symptoms of infection at S1to T1 in which case infection should be treated and the patient may after treatment be re-assessed for eligibility to enter into the study.
4. Known allergy to any of the protocol-stipulated treatment procedures, or non-tolerance of multi-layer compression therapy.
5. Ulcer which has undergone continuing high level of compression therapy for ≥12 months
6. Ulcer, which in the opinion of the Investigator is suspicious for cancer.
7. A history of more than 2 weeks' treatment with immunosuppressants (including systemic corticosteroids), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to initial screening, or treatments with such medications during the screening period, or anticipated requirement of such medications during the course of the study.
8. IGF-1 treatment or treatment with a product containing IGF-1.
9. Treatment with Pentoxifylline (Trental®) within 30-days of S1 visit.
10. Treatment with any investigational drug(s) or therapeutic device(s) within 30 days preceding screening (i.e., S1); or anticipated (patient or physician anticipates) use of any of these therapies during the course of the study.
11. Malignant disease not in remission for 5 years or more, other than basal cell carcinoma, squamous cell carcinoma of the skin or cervical carcinoma in situ, that have been successfully treated without evidence of recurrence or metastases.
12. History of radiation at the ulcer site.
13. As determined by medical history, presence of one or more medical conditions including renal, hepatic, hematologic, active auto-immune or immune diseases that, in the opinion of the Investigator, would make the patient an inappropriate candidate for this ulcer healing study.
14. Known history of having Acquired Immunodeficiency Syndrome (AIDS) or with a history of known infection with Human Immunodeficiency Virus (HIV).
15. Previous participation in any VF001-DP study within the past 6 months.
16. Ulcer has been previously treated with tissue engineered materials (e.g., Apligraf® or Dermagraft®) or other scaffold materials (e.g., Oasis®, Matristem®) within the last 30 days prior to S1.
17. Ulcer which in the opinion of the Investigator might require negative pressure ulcer therapy or hyperbaric oxygen during the course of the study.
18. New York Heart Association Class III and IV congestive heart failure, as defined by the following criteria:

    1. Class III: Symptoms with moderate exertion
    2. Class IV: Symptoms at rest
19. Uncontrolled diabetes mellitus, defined as Hemoglobin A1C >10% confirmed by the Investigator.
20. Ulcer on the dorsum of the foot or with more than 50% of the ulcer below the malleolus is excluded.
21. Known history of acromegaly.
22. Any other medical or psychological condition (including relevant laboratory abnormalities at screening) that, in the opinion of the Investigator, may suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study patient as a result of his/her participation in this clinical trial, may make patient's participation unreliable, or may interfere with study assessments. The specific justification for patients excluded under this criterion will be noted in study documents (chart notes, CRFs, etc).
23. Women unwilling to use adequate birth control, if of reproductive potential and sexually active. Adequate birth control is defined as agreement to consistently practice an effective and accepted method of contraception throughout the duration of the study.
24. Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The percentage reduction in the study ulcer area in each treatment group over the 12-week Treatment Phase. | 12-weeks
  Patient's ulcers healing rate

SECONDARY OUTCOMES:
The proportion of patients with complete study ulcer closure within the 12-week Treatment Phase | 12-weeks
  How many patient's ulcers healed?
Time to complete study ulcer closure within the 12-week Treatment Phase | 12-weeks
  Time to Ulcer Healing
Time to first instance of no study ulcer pain (i.e., pain score less than 5 mm on Visual Analog Scale [VAS]) within the 12-week Treatment Phase | 12-weeks
  Measure of pain reduction to no pain
Time to clinically meaningful study ulcer pain reduction (33% reduction on VAS) within the 12-week Treatment Phase | 12-weeks
  Measure of meaningful pain reduction
Change in Quality-of-Life metrics Euro Quality-of-Life Questionnaire EQ-5D-5L | Up to 24-weeks
  Quality of life
Change in Quality-of-Life metrics Patient Benefit Index - wound version PBI-W | Up to 24-weeks
  Quality of life - specific to chronic wounds

OTHER OUTCOMES:
The incidence of adverse events (AEs), including overall AEs, AEs related to the IP and study-ulcer-associated AEs. | Up to 24-weeks
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: William Marston, MD, Principal Investigator — UNC-Chapel Hill
Locations (16):
- United States (16):
  - ILD Research Center, Carlsbad, California
  - Limb Preservation Platform, Inc., Fresno, California
  - Alliance Research Centers, Laguna Hills, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Center for Clinical Research, Martinez, California
  - Sacramento Foot Ankle Cente, Sacramento, California
  - Bay Area Foot Care, San Francisco, California
  - NorthBay Center for Wound Care, Vacaville, California
  - University of Miami Hospital, Miami, Florida
  - Doctor Research Network (Dr Hanft), Miami, Florida
  - Miami Dade Medical Research Center (Dr Oliva), Miami, Florida
  - Spotlight Research Centre, Miami, Florida
  - Barry University School of Podiatric Medicine, North Miami Beach, Florida
  - Advanced Foot and Ankle Center, Las Vegas, Nevada
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Center for Advanced Wound Care PC, Wyomissing, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes